CLINICAL TRIAL: NCT07202728
Title: Application and Promotion of the Whole-process Management and Precision Diagnosis and Treatment System for Hydatidiform Mole: a Multi-center Cohort Study in China (CN-HM-01)
Brief Title: A Multi-center Cohort Study of Hydatidiform Mole in China (CN-HM-01)
Acronym: CN-HM-01
Status: Recruiting | Type: Observational
Sponsor: Obstetrics & Gynecology Hospital of Fudan University (Other)
Collaborators: Peking Union Medical College Hospital (Other); Shengjing Hospital (Other); Hebei Medical University Third Hospital (Other); Hainan women and children medical center (Unknown); Shenzhen Maternity & Child Healthcare Hospital (Other); Third Affiliated Hospital of Zhengzhou University (Other); Shanghai First Maternity and Infant Hospital (Other); International Peace Maternity and Child Health Hospital (Other); Shandong University (Other); First Affiliated Hospital of Zhejiang University (Other); The Affiliated Hospital of Qingdao University (Other); Gansu Provincial Maternity and Child-care Hospital/Gansu Provincial Central Hospital (Unknown); Dalian women and children's medical group (Unknown)
Responsible Party: Principal Investigator, Xin Lu, Director of Chemotherapy Unit, Gynecologic Oncology Department, Obstetrics and Gynecology Hospital,, Obstetrics & Gynecology Hospital of Fudan University
Other Study IDs: 2025-109
Record Dates: First submitted 2025-09-16; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Hydatidiform Mole
Keywords: Hydatidiform Mole; Observational Study
MeSH Terms: conditions — Hydatidiform Mole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — 1. Peripheral blood (5mL): Collected from hydatidiform mole patients in EDTA tubes for whole-genome sequencing.
  2. Uterine evacuation tissue: Selectively obtained from suspected cases for single-cell sequencing. Samples are tripartite: RNAlater (scRNA-seq), frozen (-80°C), or formalin-fixed (pathology).
  All samples are collected after obtaining informed consent, and stored under strict ethical guidelines.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hydatidiform mole: This cohort aims to support the development of evidence-based precision management strategies and facilitate nationwide promotion of optimal care practices for molar pregnancy.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This observational study aims to establish a national cohort of patients with hydatidiform mole (molar pregnancy) to investigate its malignant transformation rate and malignant transformation mechanisms, with the goal of developing and promoting precision diagnosis and treatment models across China.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically or pathologically diagnosed as hydatidiform mole.
2. Availability of complete medical records, including clinical and pathological data.
3. No evidence of myometrial invasion or metastasis.
4. Serum hCG levels normalized after uterine evacuation with at least 6 months of follow-up, OR diagnosed with postmolar gestational trophoblastic neoplasia (pGTN) during follow-up.
5. No history of psychiatric disorders, serious infectious diseases, or immune system diseases (such as systemic lupus erythematosus, myasthenia gravis, HIV infection, etc.).
6. Willing to participate in this study and sign the relevant informed consent form.

Exclusion Criteria:

1. Missing clinical data.
2. Loss to follow-up: Do not return to participating hospital for follow-up visits after uterine evacuation, or could not be contacted for subsequent monitoring of hCG changes.
3. Concomitant malignancies or autoimmune deficiency disorders (e.g., systemic lupus erythematosus, myasthenia gravis, HIV infection, etc.).
4. As determined by the investigator, the presence of medical, psychological, social, occupational, or other conditions that would violate the study protocol or impair the subject's ability to provide informed consent.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: This study will enrol women with a confirmed hydatidiform mole who have undergone uterine evacuation. Candidates must possess complete clinical and pathological records and show no myometrial invasion or distant metastasis at baseline. We will exclude those with concurrent malignancy, severe autoimmune or infectious disease, or significant psychiatric illness. Longitudinal follow-up will track malignant transformation (post-molar gestational trophoblastic neoplasia per FIGO criteria), reproductive outcomes, and health-related quality of life. By establishing a large, nationwide, multicentre cohort, we aim to clarify the epidemiology, pinpoint risk factors for malignant progression, and evaluate long-term reproductive and psychosocial outcomes in this population.
Sampling Method: Non-Probability Sample
Enrollment: 1489 (Estimated)
Dates: Start 2025-07-09 (Actual); Primary Completion 2028-08-30 (Estimated); Study Completion 2030-08-30 (Estimated)

PRIMARY OUTCOMES:
Malignant transformation of hydatidiform mole | Postoperative b-hCG levels were monitored every 1-2 weeks. While patients with PHM could discontinue follow-up after b-hCG normalization, those with CHM- given their higher risk of malignant progression- require monthly monitoring for 6 months following
  Diagnosed with pGTN according to the FIGO guideline diagnostic criteria

SECONDARY OUTCOMES:
Fertility outcomes | 1 year and 2 year
  Reproductive outcomes such as pregnancy rate, live birth rate, and miscarriage rate, following the uterine evacuation of the current molar pregnancy.
Hospital Anxiety and Depression Scale (HADS) | Pathological diagnosis, 3 months after uterine evacuation
  ordinal scale, range: 0-3, higher scores means a worse outcome
Reproductive Concerns After Cancer (RCAC) | Pathological diagnosis, 3 months after uterine evacuation
  ordinal scale, range: 1-5, higher scores mean a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Xin Lu, MD & PhD, Study Chair — Obstetrics & Gynecology Hospital of Fudan University; Yang Xiang, MD & PhD, Study Chair — Peking Union Medical College Hospital
Locations (14):
- China (14):
  - Gansu Province Maternal and Child Care Hospital, Lanzhou, Gansu
  - Shenzhen Maternity & Child Healthcare Hospital, Shenzhen, Guangdong
  - Hainan women and children medical center, Haikou, Hainan
  - Hebei Medical University Third Hospital, Shijiazhuang, Hebei
  - Third Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Dalian Women and Children medical Center, Dalian, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Center for Reproductive Medicine, Shandong University, Jinan, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Shanghai First Maternity and Infant Hospital, Shanghai, Shandong
  - Obstetrics & Gynecology Hospital of Fudan University, Shanghai, Shanghai Municipality
  - First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang
  - Peking Union Medical College Hospital, Beijing
  - International Peace Maternity and Child Health Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No